CLINICAL TRIAL: NCT03463265
Title: A Phase 2, Open-label Study of ABI-009 (Nab-Rapamycin) in Patients With Recurrent High-grade Glioma and Patients With Newly Diagnosed Glioblastoma
Brief Title: Nab-sirolimus in Recurrent High Grade Glioma and Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GBM-007
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: High Grade Recurrent Glioma and Newly Diagnosed Glioblastoma
MeSH Terms: interventions — Temozolomide; Bevacizumab; Lomustine; marizomib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A, Cohort 1: nab-sirolimus in patients with recurrent high grade glioma (Experimental): nab-Sirolimus (ABI-009, nab-rapamycin, albumin-bound rapamycin) was administered at 100 mg/m2 as a 30-minute IV infusion on Days 1 and 8 of every 21-day cycle.
  Interventions: Drug: nab-sirolimus
- Arm A, Cohort 2: nab-sirolimus + temozolomide (TMZ) in patients with recurrent high grade glioma (Experimental): nab-Sirolimus (60 mg/m 2 as a 30-minute IV infusion on Days 1, 8, and 15 of every 28-day cycle).
  Temozolomide (PO at 50 mg/m2 daily)
  Interventions: Drug: nab-sirolimus + temozolomide
- Arm A, Cohort 3: nab-sirolimus + bevacizumab in patients with recurrent high grade glioma (Experimental): nab-Sirolimus (IV 60 mg/m 2 as a 30-minute infusion on Days 1, 8, and 15 of every 28-day cycle).
  Bevacizumab (IV at a fixed dose of 5 mg/kg on Days 1 and 15 of every 28-day cycle).
  Interventions: Drug: nab-sirolimus + bevacizumab
- Arm A, Cohort 4: nab-sirolimus + lomustine (CCNU) in patients with recurrent high grade glioma (Experimental): nab-Sirolimus was administered at 60 mg/m 2 as a 30-minute IV infusion on Days 1 and 8 of every 21-day cycle.
  CCNU was administered PO at 90 mg/m2 on Day 1 of each odd 21-day cycle (ie, every 6 weeks).
  Interventions: Drug: nab-sirolimus + lomustine
- Arm A, Cohort 5: nab-sirolimus + marizomib (MRZ) in patients with recurrent high grade glioma (Experimental): nab-Sirolimus was administered at 60 mg/m 2 as a 30-minute IV infusion on Days 1, 8, and 15 of every 28-day cycle.
  MRZ was administered at 0.8 mg/m 2 as a 10-minute IV infusion on Days 1, 8, and 15 of every 28-day cycle. MRZ was administered approximately 10 minutes after the end of the nab-sirolimus infusion.
  Interventions: Drug: nab-sirolimus + marizomib (MRZ)
- Arm B: nab-sirolimus + temozolomide + radiotherapy in patients with newly diagnosed glioblastoma (Experimental): Induction Treatment (4 weeks) with nab-sirolimus (60 mg/m2 IV weekly); followed by
  Concomitant Treatment (standard of care; 2 cycles): nab-sirolimus (60 mg/m2 IV on Days 8 and 15 of every 21-day cycle) in combination with TMZ (75 mg/m2 PO daily for 6 weeks) + radiotherapy (30 × 200 cGy, 5 days/week); followed by
  Adjuvant Treatment (6 cycles) starting 4 weeks after Concomitant Treatment, with nab-sirolimus(60 mg/m2 IV on Days 1, 8, and 15 of every 28-day cycle) in combination with TMZ (150 mg/m2 PO daily on Days 1-5 of every 28-day cycle)
  Interventions: Drug: nab-sirolimus + temozolomide + radiotherapy

INTERVENTIONS:
Drug: nab-sirolimus — nab-sirolimus, single agent
  Arms: Arm A, Cohort 1: nab-sirolimus in patients with recurrent high grade glioma
Drug: nab-sirolimus + temozolomide — temozolomide, combination
  Other Names: nab-sirolimus; temozolomide
  Arms: Arm A, Cohort 2: nab-sirolimus + temozolomide (TMZ) in patients with recurrent high grade glioma
Drug: nab-sirolimus + bevacizumab — bevacizumab, combination
  Other Names: nab-sirolimus; bevacizumab
  Arms: Arm A, Cohort 3: nab-sirolimus + bevacizumab in patients with recurrent high grade glioma
Drug: nab-sirolimus + lomustine — lomustine, combination
  Other Names: nab-sirolimus; lomustine (CCNU)
  Arms: Arm A, Cohort 4: nab-sirolimus + lomustine (CCNU) in patients with recurrent high grade glioma
Drug: nab-sirolimus + marizomib (MRZ) — marizomib (MRZ), combination
  Other Names: nab-sirolimus; marizomib (MRZ)
  Arms: Arm A, Cohort 5: nab-sirolimus + marizomib (MRZ) in patients with recurrent high grade glioma
Drug: nab-sirolimus + temozolomide + radiotherapy — temozolomide + radiotherapy, combination
  Other Names: nab-sirolimus; temozolomide; radiation
  Arms: Arm B: nab-sirolimus + temozolomide + radiotherapy in patients with newly diagnosed glioblastoma

SUMMARY:
Phase 2, open-label study of nab-sirolimus in patients with recurrent high grade glioma following prior therapy and patients with newly diagnosed glioblastoma. nab-Sirolimus was administered as single agent or in combination therapies.

DETAILED DESCRIPTION:
A phase 2, open-label study of nab-sirolimus (also known as ABI-009, nab-rapamycin, albumin-bound rapamycin) in patients with recurrent high grade glioma following prior therapy and patients with newly diagnosed glioblastoma. nab-Sirolimus was administered as single agent or in combination therapies, including temozolomide, bevacizumab, lomustine, and marizomib.

ELIGIBILITY:
Inclusion Criteria Specific for Arm A

1. All subjects must have histologic evidence of high grade glioma (World Health Organization [WHO] grade 3 or grade 4) and radiographic evidence of recurrence or disease progression (defined as either a greater than 25% increase in the largest bi-dimensional product of enhancement, a new enhancing lesion, or a significant increase in T2 FLAIR). Subjects must have at least 1 measurable lesion by RANO criteria (≥ 10 mm in 2 perpendicular diameters).
2. Patients must have previously failed a treatment regimen, including radiation and/or chemotherapy.
3. No prior treatment with mTOR inhibitors.
4. No prior treatment with temozolomide for the treatment of recurrent glioma for patients entering the ABI-009 + temozolomide cohort.
5. No prior treatment with bevacizumab or any other anti-angiogenic agents, including sorafenib, sunitinib, axitinib, pazopanib, or cilengitide for the ABI-009 + bevacizumab arm.
6. No prior treatment with lomustine for the ABI-009 + lomustine arm.
7. No prior treatment with marizomib or any other proteasome inhibitors, including bortezomib, carfilzomib, or ixazomib, for patients entering the ABI-009 + marizomib cohort.
8. At least 4 weeks from surgical resection and at least 12 weeks from the end of radiotherapy prior to enrollment in this study, unless relapse is confirmed by tumor biopsy or new lesion outside of radiation field, or if there are two MRIs confirming progressive disease that are approximately 4 weeks apart.

Inclusion Criteria Specific for Arm B

1. Histologically confirmed newly diagnosed glioblastoma.
2. Patients must have had surgery and can have either non-measurable disease or a measurable post-contrast lesion after surgery detected by MRI.
3. No prior treatment with mTOR inhibitors, and no prior local or systemic therapy for GBM.

Exclusion Criteria Common for Both Arms A and B

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. Co-medication or concomitant therapy that may interfere with study results, including anti-coagulants and enzyme-inducing anti-epileptic drugs (EIAEDs).
2. History of thrombotic or hemorrhagic stroke or myocardial infarction within 6 months.
3. Pregnant or breast feeding.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics & psychiatric illness/social situations that would limit compliance with study requirements, or disorders associated with significant immunocompromised state.
5. Active gastrointestinal bleeding.
6. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥90 mm Hg.
7. Patients with history of intestinal perforations, fistula, hemorrhages and/or hemoptysis ≤6 months prior to first study treatment.
8. Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy.
9. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
10. Use of strong inhibitors and inducers of CYP3A4 within the 14 days prior to receiving the first dose of ABI-009. Additionally, use of any known CYP3A4 substrates with narrow therapeutic window (such as fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfanide) within the 14 days prior to receiving the first dose of ABI-009.
11. Known other previous/current malignancy requiring treatment within ≤ 3 years except for limited disease treated with curative intent, such as in situ prostate cancer, intracapsular renal cancer, cervical carcinoma in situ, squamous or basal cell skin carcinoma, and superficial bladder carcinoma.
12. Any comorbid condition that restricts the use of study drug and confounds the ability to interpret data from the study as judged by the Investigator or Medical Monitor.
13. Known Human Immunodeficiency Virus (HIV), or active Hepatitis B or Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - John Wayne Cancer Institute, Santa Monica, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Nab-sirolimus in Patients With Recurrent High Grade Glioma: nab-sirolimus (ABI-009, nab-rapamycin, albumin-bound rapamycin): 100 mg/m2 as a 30-minute IV infusion on Days 1 and 8 of every 21-day cycle. Two dose reduction levels allowed for toxicities: 75 mg/m2 and 60 mg/m2
- Arm A: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma: ABI-009: IV 60 mg/m 2 as a 30-minute infusion on Days 1, 8, and 15 of every 28-day cycle. If ABI-009 is well tolerated at 60 mg/m2 in the first 3 patients in the cohort, the dose may be increased to 75 mg/m2. Three dose reduction levels allowed: 45, 30, and 20 mg/m2.
  Bevacizumab: IV infusion (90 minutes 1st dose, 60 minutes 2nd dose, and 30 minutes afterward assuming tolerability) at a fixed dose of 5 mg/kg on Days 1 and 15 of every 28-day cycle. Bevacizumab administered approximately 10 minutes after the end of the ABI-009.
- Arm A: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma: ABI-009: 60 mg/m 2 as a 30-minute IV infusion on Days 1, 8, and 15 of every 28-day cycle. If ABI-009 is well tolerated at 60 mg/m2 in the first 3 patients in the cohort, the dose may be increased to 75 mg/m2. Three dose reduction levels allowed: 45, 30, and 20 mg/m2.
  Temozolomide: PO at 50 mg/m2 daily.
- Arm A: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Glioma: ABI-009: 60 mg/m 2 as a 30-minute IV infusion on Days 1 and 8 of every 21-day cycle. If ABI-009 is well tolerated at 60 mg/m2 in the first 3 patients in the cohort, the dose may be increased to 75 mg/m2. Three dose reduction levels allowed: 45, 30, and 20 mg/m2.
  Lomustine (CCNU): PO at 90 mg/m2 on Day 1 of each odd 21-day cycle (ie, every 6 weeks)
- ArmA: Nab-sirolimus + Marizomib (MRZ) in Patients With Recurrent High Grade Glioma: ABI-009: 60 mg/m 2 as a 30-minute IV infusion on Days
  1, 8, and 15 of every 28-day cycle. If ABI-009 is well tolerated at 60 mg/m2 in the first 3 patients in the cohort, the dose may be increased to 75 mg/m2. Three dose reduction levels allowed for toxicities: 45, 30, and 20 mg/m2.
  MRZ: 0.8 mg/m 2 as a 10-minute IV infusion on Days 1, 8, and 15 of every 28-day cycle. MRZ administered approximately 10 minutes after the end of the ABI-009 infusion.
- Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma: Concomitant Treatment: starting 1 week after the completion of Induction Treatment and lasting for 6 weeks (2 cycles).
  ABI-009: IV at 60 mg/m2 as a 30-minute IV infusion on Days 8 and 15 of every 21-day cycle. Three dose reduction levels allowed: 45, 30, and 20 mg/m2.
  Temozolomide: 75 mg/m2 PO daily for 6 weeks. Focal RT: daily at 30 x 200 cGy, 5 days/week for a total dose of 60 Gy (or equivalent regimens as per RTOG guidelines)
Period: Overall Study
Arm/Group | Arm A: Nab-sirolimus in Patients With Recurrent High Grade Glioma | Arm A: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma | Arm A: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma | Arm A: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Glioma | ArmA: Nab-sirolimus + Marizomib (MRZ) in Patients With Recurrent High Grade Glioma | Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma
Started | 7 | 6 | 9 | 4 | 10 | 26
Completed | 7 | 6 | 9 | 4 | 10 | 26
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nab-sirolimus in Patients With Recurrent High Grade Glioma | Arm A: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma | Arm A: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma | Arm A: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Glioma | ArmA: Nab-sirolimus + Marizomib (MRZ) in Patients With Recurrent High Grade Glioma | Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma | Total
Number analyzed (Participants) | 7 | 6 | 9 | 4 | 10 | 26 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 7 | 4 | 9 | 13 | 42
  >=65 years | 2 | 2 | 2 | 0 | 1 | 13 | 20
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 78] | 53.5 [34 to 71] | 60 [45 to 70] | 53 [38 to 59] | 52.5 [27 to 72] | 64 [27 to 80] | 60 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 3 | 6 | 15
  Male | 5 | 4 | 8 | 3 | 7 | 20 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 3 | 0 | 3 | 3 | 13
  Not Hispanic or Latino | 6 | 2 | 6 | 4 | 7 | 23 | 48
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 6 | 9 | 4 | 9 | 25 | 58
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 9 | 4 | 10 | 26 | 62

OUTCOME MEASURES:

1. Primary Outcome: ORR
Description: Objective overall response rate (ORR, according to Response Assessment in Neuro-Oncology [RANO]) by investigator-assessed radiologic review and defined as the proportion of patients who achieved a confirmed partial response (PR) or confirmed complete response (CR) per RANO 2010 criteria. PR is defined as greater than or equal to 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks.
Time Frame: Through study completion (up to 48 months)
Population: Efficacy Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Arm A, Cohort 1: Nab-sirolimus in Patients With Recurrent High Grade Glioma: nab-Sirolimus single agent (100 mg/m2 as a 30-minute IV infusion on Days 1 and 8 of every 21-day cycle)
- Arm A, Cohort 2: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma: nab-Sirolimus (60 mg/m 2 as a 30-minute IV infusion on Days 1, 8, and 15 of every 28-day cycle) plus Temozolomide (PO at 50 mg/m2 daily)
- Arm A, Cohort 3: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma: nab-Sirolimus (IV 60 mg/m 2 as a 30-minute infusion on Days 1, 8, and 15 of every 28-day cycle) plus Bevacizumab (IV at a fixed dose of 5 mg/kg on Days 1 and 15 of every 28-day cycle)
- Arm A, Cohort 4: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Glioma: nab-Sirolimus (60 mg/m 2 as a 30-minute IV infusion on Days 1 and 8 of every 21-day cycle) plus Lomustine (CCNU, PO at 90 mg/m2 on Day 1 of each odd 21-day cycle, ie, every 6 weeks)
- Arm A, Cohort 5: Nab-sirolimus + Marizomib in Patients With Recurrent High Grade Glioma: nab-Sirolimus (60 mg/m 2 as a 30-minute IV infusion on Days 1, 8, and 15 of every 28-day cycle) plus Marizomib (0.8 mg/m 2 as a 10-minute IV infusion on Days 1, 8, and 15 of every 28-day cycle)
- Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma: 4-week Induction Treatment with nab-sirolimus followed by Concomitant Treatment of nab-sirolimus + temozolomide + RT for 2 cycles, followed by adjuvant treatment of nab-sirolimus + temozolomide for 6 cycles
Arm/Group | Arm A, Cohort 1: Nab-sirolimus in Patients With Recurrent High Grade Glioma | Arm A, Cohort 2: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma | Arm A, Cohort 3: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma | Arm A, Cohort 4: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Glioma | Arm A, Cohort 5: Nab-sirolimus + Marizomib in Patients With Recurrent High Grade Glioma | Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 10 | 26
percentage of patients | 0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 11.5 [2.4 to 30.2]

2. Secondary Outcome: Median PFS
Description: Progression-free Survival defined as number of months from the date of the first dose of study drug to the first observation of a disease progression or death due to any cause.
  Progression is assessed according to Response Assessment in Neuro-Oncology (RANO) 2010 criteria based on MRI imaging, and includes ≥25% increase in the sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids.
Time Frame: Through study completion (up to 48 months)
Population: Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A, Cohort 1: Nab-sirolimus in Patients With Recurrent High Grade Glioma | Arm A, Cohort 2: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma | Arm A, Cohort 3: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma | Arm A, Cohort 4: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Glioma | Arm A, Cohort 5: Nab-sirolimus + Marizomib in Patients With Recurrent High Grade Glioma | Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 10 | 26
months | 1.7 [1.3 to NA] — Upper limit was not reached due to insufficient number of participants with events | 11.3 [5.2 to NA] — Upper limit was not reached due to insufficient number of participants with events | 3.1 [1.7 to 9.2] | 3.8 [1.4 to NA] — Upper limit was not reached due to insufficient number of participants with events | 1.7 [0.9 to 3.5] | 7.5 [6.2 to 14.4]

3. Secondary Outcome: PFS Rate at 6 Months and 12 Months
Description: Progression-free survival rate at 6 months and 12 months was calculated as the proportion of patients who were progression-free and alive at 6 and 12 months, respectively.
  Progression is assessed according to Response Assessment in Neuro-Oncology (RANO) 2010 criteria based on MRI imaging, and includes ≥25% increase in the sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids.
Time Frame: 6 and 12 months
Population: Efficacy Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A, Cohort 1: Nab-sirolimus in Patients With Recurrent High Grade Glioma | Arm A, Cohort 2: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma | Arm A, Cohort 3: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma | Arm A, Cohort 4: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Glioma | Arm A, Cohort 5: Nab-sirolimus + Marizomib in Patients With Recurrent High Grade Glioma | Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 10 | 26
percentage of patients
  PFS at 6 months | 0.0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 75.0 [12.8 to 96.1] | 37.5 [8.7 to 67.4] | 25.0 [0.9 to 66.5] | 10.0 [0.6 to 35.8] | 76.9 [55.7 to 88.9]
  PFS at 12 months | 0.0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 50.0 [5.8 to 84.5] | 12.5 [0.7 to 42.3] | 0.0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 0.0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 36.4 [18.5 to 54.7]

4. Secondary Outcome: OS
Description: Median Overall Survival
Time Frame: Through study completion (up to 48 months)
Population: Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A, Cohort 4: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Gliom: nab-Sirolimus (60 mg/m 2 as a 30-minute IV infusion on Days 1 and 8 of every 21-day cycle) plus Lomustine (CCNU, PO at 90 mg/m2 on Day 1 of each odd 21-day cycle, ie, every 6 weeks)
Arm/Group | Arm A, Cohort 1: Nab-sirolimus in Patients With Recurrent High Grade Glioma | Arm A, Cohort 2: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma | Arm A, Cohort 3: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma | Arm A, Cohort 4: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Gliom | Arm A, Cohort 5: Nab-sirolimus + Marizomib in Patients With Recurrent High Grade Glioma | Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 10 | 26
months | 7.2 [2.7 to NA] — Upper limit was not reached due to insufficient number of participants with events | 13.8 [5.2 to NA] — Upper limit was not reached due to insufficient number of participants with events | 6.8 [1.7 to 13.1] | 7.5 [5.4 to NA] — Upper limit was not reached due to insufficient number of participants with events | 6.7 [1.7 to 9.2] | 13.3 [7.9 to 23.2]

5. Secondary Outcome: OS at 12 Months
Description: Overall Survival rate at 12 months
Time Frame: 12 months
Population: Efficacy Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A, Cohort 1: Nab-sirolimus in Patients With Recurrent High Grade Glioma | Arm A, Cohort 2: Nab-sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma | Arm A, Cohort 3: Nab-sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma | Arm A, Cohort 4: Nab-sirolimus + Lomustine in Patients With Recurrent High Grade Glioma | Arm A, Cohort 5: Nab-sirolimus + Marizomib in Patients With Recurrent High Grade Glioma | Arm B: Nab-sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 10 | 26
percentage of patients | 0.0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 66.7 [19.5 to 90.4] | 25.0 [3.7 to 55.8] | 25.0 [0.9 to 66.5] | 0.0 [NA to NA] — The 95% CI could not be calculated as there were no patients with an event. | 53.8 [33.3 to 70.6]

ADVERSE EVENTS:
Time Frame: Safety and tolerability were monitored through continuous reporting of treatment-emergent and treatment-related adverse events (AEs) and serious AEs, from the time the patient signed informed consent until 28 days after the last dose of nab-sirolimus, for up to 48 months (study duration).
Description: All patients were evaluated for safety analysis if they received at least one dose of nab-sirolimus. Treatment with nab-sirolimus continued until disease progression or unacceptable AEs. Safety and tolerability was monitored during treatment (from signing of informed consent till 28 days after last dose), through reporting of AEs, serious AEs, laboratory abnormalities, and incidence of dose modifications, dose delay/dose not given, and/or premature discontinuation of nab-sirolimus due to an AE.
Arm/Group | Arm A, Cohort 1: Nab-Sirolimus in Patients With Recurrent High Grade Glioma | Arm A, Cohort 2: Nab-Sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma | Arm A, Cohort 3: Nab-Sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma | Arm A, Cohort 4: Nab-Sirolimus + Lomustine in Patients With Recurrent High Grade Glioma | Arm A, Cohort 5: Nab-Sirolimus + Marizomib in Patients With Recurrent High Grade Glioma | Arm B: Nab-Sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma
All-Cause Mortality (participants affected / at risk) | 7/7 | 4/6 | 8/9 | 4/4 | 10/10 | 19/26
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/9 | 1/4 | 0/10 | 1/26
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 8/9 | 4/4 | 10/10 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, Cohort 1: Nab-Sirolimus in Patients With Recurrent High Grade Glioma (N=7) | Arm A, Cohort 2: Nab-Sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma (N=6) | Arm A, Cohort 3: Nab-Sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma (N=9) | Arm A, Cohort 4: Nab-Sirolimus + Lomustine in Patients With Recurrent High Grade Glioma (N=4) | Arm A, Cohort 5: Nab-Sirolimus + Marizomib in Patients With Recurrent High Grade Glioma (N=10) | Arm B: Nab-Sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma (N=26)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myelosuppression (thrombocytopenia) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myelossupression (neutropenia) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, Cohort 1: Nab-Sirolimus in Patients With Recurrent High Grade Glioma (N=7) | Arm A, Cohort 2: Nab-Sirolimus + Temozolomide in Patients With Recurrent High Grade Glioma (N=6) | Arm A, Cohort 3: Nab-Sirolimus + Bevacizumab in Patients With Recurrent High Grade Glioma (N=9) | Arm A, Cohort 4: Nab-Sirolimus + Lomustine in Patients With Recurrent High Grade Glioma (N=4) | Arm A, Cohort 5: Nab-Sirolimus + Marizomib in Patients With Recurrent High Grade Glioma (N=10) | Arm B: Nab-Sirolimus + Temozolomide + Radiotherapy in Patients With Newly Diagnosed Glioblastoma (N=26)
Mucositis (Gastrointestinal disorders) | 4 | 5 | 2 | 2 | 1 | 14
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 4 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 1
Myelosuppression (thrombocytopenia) (Blood and lymphatic system disorders) | 2 | 3 | 5 | 3 | 7 | 14
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 3
Myelosuppression (anemia) (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 3 | 3 | 3 | 12
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1 | 2 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 6
Myelossupression (neutropenia) (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 3
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 2 | 2 | 3 | 2 | 2 | 9
Mucosal inflammation (General disorders) | 0 | 0 | 3 | 0 | 0 | 6
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 1
ALT (Investigations) | 0 | 2 | 2 | 0 | 0 | 4
AST (Investigations) | 0 | 1 | 2 | 0 | 0 | 4
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 3
Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03463265/Prot_SAP_001.pdf